CLINICAL TRIAL: NCT04385979
Title: Comparison of Curcumin and NanoCurcumin in Recurrent Aphthous Stomatitis
Brief Title: Curcumin and Nanocurcumin in Oral Aphthous Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahin Bakhshi, Associate Professor, Shahid Beheshti University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBMU1
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Recurrent Aphthous Ulcer; Recurrent Aphthous Stomatitis
Keywords: Recurrent Aphthous Stomatitis; Curcumin; Nanocurcumin; management
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin (Active Comparator): %2 Curcumin gel
  Interventions: Other: Gel
- Nanocurcumin (Active Comparator): %1 NanoCurcumin gel
  Interventions: Other: Gel

INTERVENTIONS:
Other: Gel — containing herbal Curcumin or NanoCurcumin

SUMMARY:
Recurrent aphthous ulcer is a painful inflammatory lesion with a high prevalence. Since the etiology is not clear, several strategies have been proposed to reduce pain and severity of its symptoms. Today, curcumin is considered as an herbal medicine with anti-inflammatory properties. Treatment or control of various inflammatory diseases has been proposed, but its low solubility in water has reduced bioavailability, while the use of nanoparticle pharmaceutical techniques has been able to solve these problems. Therefore, the aim of the present study was to evaluate the clinical efficacy of a new topical curcumin gel with nano-technology and compare it with 2% curcumin gel in patients with recurrent aphthous ulcers.

This randomized clinical trial was performed on 48 patients assigned to two groups (nano-curcumin gel) and (curcumin gel). Before treatment, the size of the wound and VAS were measured. After intervention, the two variables were measured again on the fourth and seventh days , then the amount of improvement was quantitatively and qualitatively compared in the two groups and a significant level of less than 0.05 was considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with minor and recurrent aphthous ulcer lesions within 48 hours and Aphthous like Lesions

Exclusion Criteria:

* Wounds are in inaccessible areas (such as posterior palate). If a person suffers from systemic disease (through questioning the patient) Patients with turmeric allergy and any type of gel used in this study. Pregnant or lactating women .. accompany with other mucosal lesions. Do not take any other medicine while taking intervention Major or herpeti form of aphthous ulcer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Wound size | one week
  The ulcer size was evaluated by determining the distance between two opposed boundaries of the ulcer edge, using a periodontal probe in millimeters.
Pain score | one week
  Pain assessment scale, visual analog scale (VAS) comprising of a 10-cm straight line among ends, with 0 representing no pain (better outcome) and 10 for intolerable pain (worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Mahinbakhshi@Sbmu.Ac.Ir, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided